CLINICAL TRIAL: NCT01273974
Title: The Comparison of Serum Antibody Response to Standard Intramuscular and Half Dose Intradermal Influenza Vaccine in Hemodialysis Patients in Shiraz City in 1388.
Brief Title: The Immunogenicity of Intradermal Influenza Vaccination in Hemodialysis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 89-5905
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-08

CONDITIONS: Hemodialysis Patients
Keywords: intradermal influenza vaccine; hemodialysis patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intradermal influenza vaccine (Experimental)
  Interventions: Biological: intradermal influenza vaccine
- intramuscular influenza vaccine (Active Comparator)
  Interventions: Biological: intramuscular influenza vaccine

INTERVENTIONS:
Biological: intradermal influenza vaccine — 0.25ml ,intradermal
  Arms: intradermal influenza vaccine
Biological: intramuscular influenza vaccine — 0.5ml,intramuscular
  Arms: intramuscular influenza vaccine

SUMMARY:
The purpose of this study is to determine whether half-dose intradermal influenza vaccine is as immunogenic as standard dose intramuscular vaccine in hemodialysis patients.

DETAILED DESCRIPTION:
Hemodialysis patients are at high risk of influenza infection due to suppress immune status.It is recommended to immunize them against influenza annually.in intradermal vaccination antigens directly present to the large numbers of antigen-presenting cells in the skin and it may cause greater immunogenicity than in the intramuscular method. Reduced-dose intradermal influenza vaccine is immunogenic in healthy adult, patients with solid cancer and three groups of immunocompromized patients including Rheumatologic patients treated with anti-TNF, HIV-infected and stem cell transplanted patients.

In this study we compare the efficacy of influenza vaccines in half dose intradermal and standard intramuscular methods among hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients under chronic hemodialysis

Exclusion Criteria:

* history of flu infection in last month
* history of flu vaccination in 2009
* hospitalization in last month
* taking immune suppressants drugs
* hemodialysis less than twice weekly

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
vaccine effectiveness | 3 months
  serum antibody response measured by ELIZA method time frame:1 and 3 months after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad mahdi Sagheb, Principal Investigator — Shiraz University Of Medical Science; Samira Saeian, Principal Investigator — Shiraz University Of Medical Science; Jamshid Roozbeh, Principal Investigator — Shiraz University Of Medical Science
Locations (1):
- Shiraz University Of Medical Science, Shiraz, Iran